CLINICAL TRIAL: NCT06147128
Title: Proficiency Based Progression Training Versus Traditional Training During a Robotic Emergency Conversion Due to a Vessel Injury in a Simulated Setting: a Prospective, Randomized, Multicenter Clinical Trial: The T-REC Trial
Brief Title: PBP vs Traditional Training: the T-REC Trial
Acronym: T-REC
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Orsi Academy (Other)
Responsible Party: Sponsor
Other Study IDs: T-REC
Record Dates: First submitted 2023-11-19; First posted 2023-11-27 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Educational Problems
Keywords: Training; Robotic surgery; Proficiency based progression; Emergency undocking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Active Comparator: Traditional Trained: Trainees in the Traditional trained group will have an e-learning didactic component (specifically on the steps of the procedure, clinical aspects of the procedure, published evidence etc) which they must complete before training by a procedure expert. On completion of the e-learning module the trainees will complete a summative assessment of their knowledge. The trainees will then be shown how and then trained to perform an emergency scenario where open conversion is necessary due to vessel injury during robotic surgery task. The scenario will be demonstrated initially by an expert and who will then proctor the trainees in the same technique.
  Interventions: Procedure: Emergency scenario in a simulated setting where open conversion is necessary due to vessel injury during robotic surgery on a dry lab model
- Experimental: PBP for Technical emergency undocking skills: Participants in the PBP trained group will follow the exact same e-learning didactic course as the Traditional trained group but the PBP group will be required to pass a test of procedure knowledge on TS before continuing to the robotic surgical training element. The trainees knowledge will be assessed in a formative and summative fashion. After the trainees initial assessment, procedure-specific and validated procedure metrics will be used to teach them the steps of the emergency undocking procedure, as well as the correct (and incorrect) way to perform it. The metrics will be used to give to the trainees performance feedback with specific advice on how they might improve their performance, in the regards of technical skills.
  Interventions: Procedure: Emergency scenario in a simulated setting where open conversion is necessary due to vessel injury during robotic surgery on a dry lab model
- Experimental: PBP for Non-Technical emergency undocking skills: Participants in the PBP trained group will follow the exact same e-learning didactic course as the Traditional trained group but the PBP group will be required to pass a test of procedure knowledge on NTS before continuing to the robotic surgical training element. The trainees knowledge will be assessed in a formative and summative fashion. After the trainees initial assessment, procedure-specific and validated procedure metrics will be used to teach them the steps of the emergency undocking procedure, as well as the correct (and incorrect) way to perform it. The metrics will be used to give to the trainees performance feedback with specific advice on how they might improve their performance, in the regards of non-technical skills.
  Interventions: Procedure: Emergency scenario in a simulated setting where open conversion is necessary due to vessel injury during robotic surgery on a dry lab model
- Experimental: PBP for Technical and Non-Technical emergency undocking skills: Participants in the PBP trained group will follow the exact same e-learning didactic course as the Traditional trained group but the PBP group will be required to pass a test of procedure knowledge on both TS and NTS before continuing to the robotic surgical training element. The trainees knowledge will be assessed in a formative and summative fashion. After the trainees initial assessment, procedure-specific and validated procedure metrics will be used to teach them the steps of the emergency undocking procedure, as well as the correct (and incorrect) way to perform it. The metrics will be used to give to the trainees performance feedback with specific advice on how they might improve their performance, in the regards of technical and non-technical skills.
  Interventions: Procedure: Emergency scenario in a simulated setting where open conversion is necessary due to vessel injury during robotic surgery on a dry lab model

INTERVENTIONS:
Procedure: Emergency scenario in a simulated setting where open conversion is necessary due to vessel injury during robotic surgery on a dry lab model — Performance of emergency scenario where open conversion is necessary due to vessel injury during robotic surgery on a dry lab model with Da Vinci robotic system
  Other Names: Robotic emergency conversion

SUMMARY:
This randomized controlled trial aims to compare the effectiveness of traditional training approach to training with the proficiency-based progression (PBP) approach for teaching the technical skills (TS) and non-technical skills (NTS) for surgeons in the context of an emergency scenario where open conversion is necessary due to vessel injury during robotic surgery.

DETAILED DESCRIPTION:
In a prospective, randomized and blinded study surgical residents (n = 48) from Belgium university (i.e. the Katholieke Universiteit [KU] Leuven and University of Gent residency training programs) will be enrolled and randomized to Traditional type training proficiency-based progression (PBP) training to learn how to perform an emergency scenario where open conversion is necessary due to vessel injury during robotic surgery on a dry lab model. Specifically, this study will include four independent arms, each employing different training methodologies for technical skills (TS) and non-technical skills (NTS).

Group 1 will receive standard training for both TS and NTS. Group 2 will receive PBP training for TS and standard training for NTS. Group 3 will receive standard training for TS and PBP training for NTS. Group 4 will receive PBP training for both TS and NTS.

All four group will receive the same e-learning on TS and NTS (on an emergency scenario where (simulated) open conversion is necessary due to vessel injury during robotic surgery on a dry lab model). The PBP trained group will however be required to demonstrate quantitively defined proficiency benchmarks for training progression (i.e., for the e-learning, TS and NTS). The Traditional trained group will train in the same laboratory for a case-matched period of time as the PBP group, with the same level of supervising faculty proctors and using the same training resources but with no proficiency benchmarks.

Investigators will be trained in pairs to assess performance from a pre-defined set of explicitly defined binary metric events reliably (inter-rater reliability > 0.8). They will also be blinded as to the identity of the trainee performing the procedure, how they were trained (i.e., group) and procedure order.

H1 It is hypothesized that implementation of PBP training in teaching TS and NTS for surgeons in the context of an emergency scenario where (simulated) open conversion is necessary due to vessel injury during robotic surgery, leads to better surgical training outcomes (i.e., lower number of performance errors) when compared to traditional training.

ELIGIBILITY:
Inclusion Criteria:

* recently accepted, form first to last year residents' gynecology and obstetrics, urology and general surgery.
* Ability to perform a laparotomy

Exclusion Criteria:

* Any robotic experience with emergency undocking.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents in urology, surgery and gynecology from Belgium universities (i.e. the KU Leuven and University of Gent residency training programs) from the first to the last year.
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2023-12-03 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Comparison between PBP training versus traditional training for an emergency scenario where an open conversion is necessary due to a (simulated) vessel injury during robotic surgery on a dry lab model with Da Vinci robotic system. | 1 year
  Proficiency level will be determined by objectively assessed, validated, binary performance operative metrics where the proficiency benchmark is defined on the mean of the objectively assessed performance of experienced practitioners.
  The aim of this study is to report the main performance outcomes of the T-REC trial. The investigators will compare differences between four groups in performance level as assessed by binary performance metrics of an emergency scenario where open conversion is necessary due to vessel injury during robotic surgery on a dry lab model with Da Vinci robotic system.
  The four groups deffers for the training methodology used (PBP vs traditional training). The dependant variables will be the i) time required to complete the procedure, ii) the number of procedure steps completed, iii) the number of errors made, iv) the number of critical errors made and whether the procedure was completed or not.

SECONDARY OUTCOMES:
Trainee's satisfaction as assessed by questionnaire. Does it influence outcome of surgical training? Comparison between PBP training versus traditional training group. | 2 years
  Satisfaction of a surgical trainee is often thought to be key for training quality and a predictor of good outcome of surgical training. At the end of the T-REC trial, all participants were asked to complete an online questionnaire where their satisfaction with the adopted training method was asked for using a Likert scale.
  Hypothesis is that trainee's satisfaction does NOT correlate with training outcome and that satisfaction is NOT a good determinator of training quality.
Correlation between live and video-based scoring of surgical performance | 2 years
  Surgical performance is often assessed live during surgery. However, one might miss specific details of performance. A possible answer to this query lies in video-based scoring of a surgical task. However, does video-based scoring reflects the same surgical quality? Moreover, one could question the ethical aspect of non-live scoring of surgical performance.
  In the T-REC trial, all surgical tasks were scored live and video-based afterwards. The correlation in metrics-based performance scores between live and video-based assessment will be investigated.
  Hypothesis is that there will be no differences. The investigators will try to answer the question which scoring method will give the trainee the highest chance of reaching proficiency?
Reporting the outcome of the e-learning scores from an online proficiency questionnaire on an online learning platform. | 2 years
  During the T-REC trial, all participants will be required to complete an online assessment. This will done on an online learning platform. A proficiency benchmark will be defined based on the mean score of experts on the same assessment. The PBP group will be required to pass this assessment in order to move forward to the clinical training in the lab. The Control group will be required to complete the exact same online assessment before and after their training and after performing the final task. The investigators aim to do a comparison between proficiency based progression training versus traditional training for a emergency scenario where open conversion is necessary due to vessel injury during robotic surgery on a dry lab model with Da Vinci robotic system task in the regard of the e-learning scores.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Collà Ruvolo, MD, Principal Investigator — Orsi Academy
Locations (1):
- Orsi Academy, Melle, Oost - Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pellegrini CA. Surgical education in the United States: navigating the white waters. Ann Surg. 2006 Sep;244(3):335-42. doi: 10.1097/01.sla.0000234800.08200.6c. No abstract available. PMID 16926559
- [Result] Cuschieri A. Whither minimal access surgery: tribulations and expectations. Am J Surg. 1995 Jan;169(1):9-19. doi: 10.1016/s0002-9610(99)80104-4. No abstract available. PMID 7818004
- [Result] Gallagher AG. Metric-based simulation training to proficiency in medical education:- what it is and how to do it. Ulster Med J. 2012 Sep;81(3):107-13. PMID 23620606
- [Result] Gallagher AG, Ritter EM, Champion H, Higgins G, Fried MP, Moses G, Smith CD, Satava RM. Virtual reality simulation for the operating room: proficiency-based training as a paradigm shift in surgical skills training. Ann Surg. 2005 Feb;241(2):364-72. doi: 10.1097/01.sla.0000151982.85062.80. PMID 15650649
- [Result] Breen D, O'Brien S, McCarthy N, Gallagher A, Walshe N. Effect of a proficiency-based progression simulation programme on clinical communication for the deteriorating patient: a randomised controlled trial. BMJ Open. 2019 Jul 9;9(7):e025992. doi: 10.1136/bmjopen-2018-025992. PMID 31289064
- [Result] Kallidaikurichi Srinivasan K, Gallagher A, O'Brien N, Sudir V, Barrett N, O'Connor R, Holt F, Lee P, O'Donnell B, Shorten G. Proficiency-based progression training: an 'end to end' model for decreasing error applied to achievement of effective epidural analgesia during labour: a randomised control study. BMJ Open. 2018 Oct 15;8(10):e020099. doi: 10.1136/bmjopen-2017-020099. PMID 30327396
- [Result] Cates CU, Lonn L, Gallagher AG. Prospective, randomised and blinded comparison of proficiency-based progression full-physics virtual reality simulator training versus invasive vascular experience for learning carotid artery angiography by very experienced operators. BMJ Simul Technol Enhanc Learn. 2016 Feb 8;2(1):1-5. doi: 10.1136/bmjstel-2015-000090. eCollection 2016. PMID 35516451
- [Result] Angelo RL, Ryu RK, Pedowitz RA, Beach W, Burns J, Dodds J, Field L, Getelman M, Hobgood R, McIntyre L, Gallagher AG. A Proficiency-Based Progression Training Curriculum Coupled With a Model Simulator Results in the Acquisition of a Superior Arthroscopic Bankart Skill Set. Arthroscopy. 2015 Oct;31(10):1854-71. doi: 10.1016/j.arthro.2015.07.001. Epub 2015 Sep 2. PMID 26341047
- [Result] Van Sickle KR, Ritter EM, Baghai M, Goldenberg AE, Huang IP, Gallagher AG, Smith CD. Prospective, randomized, double-blind trial of curriculum-based training for intracorporeal suturing and knot tying. J Am Coll Surg. 2008 Oct;207(4):560-8. doi: 10.1016/j.jamcollsurg.2008.05.007. Epub 2008 Jul 14. PMID 18926460
- [Result] Ahlberg G, Enochsson L, Gallagher AG, Hedman L, Hogman C, McClusky DA 3rd, Ramel S, Smith CD, Arvidsson D. Proficiency-based virtual reality training significantly reduces the error rate for residents during their first 10 laparoscopic cholecystectomies. Am J Surg. 2007 Jun;193(6):797-804. doi: 10.1016/j.amjsurg.2006.06.050. PMID 17512301
- [Result] Seymour NE, Gallagher AG, Roman SA, O'Brien MK, Bansal VK, Andersen DK, Satava RM. Virtual reality training improves operating room performance: results of a randomized, double-blinded study. Ann Surg. 2002 Oct;236(4):458-63; discussion 463-4. doi: 10.1097/00000658-200210000-00008. PMID 12368674
- [Result] de Vries EN, Ramrattan MA, Smorenburg SM, Gouma DJ, Boermeester MA. The incidence and nature of in-hospital adverse events: a systematic review. Qual Saf Health Care. 2008 Jun;17(3):216-23. doi: 10.1136/qshc.2007.023622. PMID 18519629
- [Result] Gawande AA, Zinner MJ, Studdert DM, Brennan TA. Analysis of errors reported by surgeons at three teaching hospitals. Surgery. 2003 Jun;133(6):614-21. doi: 10.1067/msy.2003.169. PMID 12796727
- [Result] Greenberg CC, Regenbogen SE, Studdert DM, Lipsitz SR, Rogers SO, Zinner MJ, Gawande AA. Patterns of communication breakdowns resulting in injury to surgical patients. J Am Coll Surg. 2007 Apr;204(4):533-40. doi: 10.1016/j.jamcollsurg.2007.01.010. PMID 17382211
- [Result] Collins JW, Dell'Oglio P, Hung AJ, Brook NR. The Importance of Technical and Non-technical Skills in Robotic Surgery Training. Eur Urol Focus. 2018 Sep;4(5):674-676. doi: 10.1016/j.euf.2018.08.018. Epub 2018 Sep 11. PMID 30217631
- [Result] Mazzone E, Puliatti S, Amato M, Bunting B, Rocco B, Montorsi F, Mottrie A, Gallagher AG. A Systematic Review and Meta-analysis on the Impact of Proficiency-based Progression Simulation Training on Performance Outcomes. Ann Surg. 2021 Aug 1;274(2):281-289. doi: 10.1097/SLA.0000000000004650. PMID 33630473
- See also: Gallagher Anthony, O'Sullivan Gerarld. Fundamentals of Surgical Simulation [Internet]. London: Springer London; 2012 — http://link.springer.com/10.1007/978-0-85729-763-1